CLINICAL TRIAL: NCT02357290
Title: Open-Label Study of N-Acetylcysteine in Children and Adolescents Ages 5-17 With Bipolar I, Bipolar II, and Bipolar Spectrum Disorder
Brief Title: Open-Label Study of N-Acetylcysteine in Children and Adolescents 5-17 With Bipolar Spectrum Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Janet Wozniak, MD, Associate Professor of Psychiatry, Harvard Medical School; Medical Director, Child and Adolescent Outpatient Psychiatry Services; Director, Pediatric Bipolar Clinical and Research Program in Pediatric Psychopharmacology, Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014P002011
Record Dates: First submitted 2015-02-02; First posted 2015-02-06 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Bipolar Disorder
Keywords: mania; temper tantrum; irritability; mood; bipolar
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label Treatment with NAC (Experimental): 12-week, open-label treatment with NAC. Subjects will be treated with the following dose:
  Subjects ages 5-12:
  Week 1: 900mg po daily Weeks 2+: 900mg po QAM, 900mg po QPM
  Subjects ages 13-17:
  Week 1: 900mg po daily Weeks 2-3: 900mg po QAM, 900mg po QPM Weeks 4+: 1800mg po QAM, 900mg po QPM
  In Weeks 3-12 for subjects ages 13-17, we will encourage twice per day dosing, but we will permit daily dosing if needed for adherence.
  Interventions: Drug: Open-label Treatment with N-Acetylcysteine

INTERVENTIONS:
Drug: Open-label Treatment with N-Acetylcysteine

SUMMARY:
Children between the ages of 5-17 years old who have or display symptoms of emotional dysregulation (explosiveness, mood swings, irritability, and/or violent behavior) are invited to participate in a 12-week research study to determine the effectiveness and safety of the natural treatment N-acetylcysteine (NAC) for children with emotional and behavioral problems. After undergoing a comprehensive evaluation by medical doctors with a specialty in this area, children who are found eligible to participate in this research study will be treated with NAC. Following the evaluation period, this research study requires 12 weekly visits, either in our office or over the phone, in an effort to closely monitor each child's response to the medication. Eligible participants will receive study-related evaluations and weekly study visits with our study doctors at no cost.

DETAILED DESCRIPTION:
This will be a 12-week, open-label study of NAC in the treatment of bipolar disorder in children and adolescents. Subjects will include youth ages 5-17 years with a bipolar spectrum disorder (type I, II, or NOS), mixed, manic, or hypomanic state, according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition DSM-5 (American Psychiatric Association, 2013). The primary outcome measures will be improvement in manic symptoms as measured by the Young Mania Rating Scale (YMRS) and improvement in depressive symptoms as measured by the Child Depression Rating Scale (CDRS).

Bipolar diagnoses will be made according to the DSM-5 in a clinical evaluation by a Child Psychiatrist and confirmed using the Schedule for Affective Disorders and Schizophrenia for School-Age Children - Epidemiological Version (K-SADS-E)(Orvaschel, 1994). All subjects must have a YMRS score of at least 15. Only patients who are not responding to their current treatment regimen will be tapered from their medications; youth on concomitant psychiatric medications will be permitted to continue those medications as listed in the concomitant medication section.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 5-17 years of age
* Subjects must have a DSM-IV diagnosis of a bipolar spectrum disorder (type I, II, or Not Otherwise Specified) and currently display mixed, manic, or hypomanic symptoms (without psychotic features) according to clinical assessment based on the DSM-IV and confirmed with structured diagnostic interview
* Subjects and their legal representative must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator and to cooperate with all tests and examinations required by the protocol
* Subjects and their legal representatives must be considered reliable.
* Each subject and his/her authorized legal representative must understand the nature of the study. The subject's authorized legal representative must provide written consent and the subject must provide written assent.
* Subjects must have an initial score on the YMRS of at least 15.

Exclusion Criteria:

* Investigator and his/her immediate family (defined as the investigator's spouse, parent, child, grandparent, or grandchild)
* Serious or unstable illness including hepatic, rental, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease
* Uncorrected hypothyroidism or hyperthyroidism
* History of sensitivity to N-acetylcysteine, a history of intolerance to N-acetylcysteine, or a non-responder after 2 months of treatment at adequate doses as determined by the clinician
* Severe allergies or multiple adverse drug reactions
* Current or past history of seizures
* Active substance abusers, per clinician judgment
* Judged clinically to be at serious suicidal risk
* Current diagnosis of schizophrenia
* Pregnancy
* C-SSRS score ≥ 4
* IQ < 70

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Wozniak, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wozniak J, DiSalvo M, Farrell A, Vaudreuil C, Uchida M, Ceranoglu TA, Joshi G, Cook E, Faraone SV, Biederman J. Findings from a pilot open-label trial of N-acetylcysteine for the treatment of pediatric mania and hypomania. BMC Psychiatry. 2022 May 3;22(1):314. doi: 10.1186/s12888-022-03943-x. PMID 35505312

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-Label Treatment With NAC: 12-week, open-label treatment with NAC.
Period: Overall Study
Arm/Group | Open-Label Treatment With NAC
Started | 40
Exposed | 26
Completed | 14
Not Completed | 26

BASELINE CHARACTERISTICS:
Population: Analysis was only conducted for subjects exposed to study treatment for at least 2 weeks.
Arm/Group | Open-Label Treatment With NAC
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.0 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 19
  More than one race | 2
  Unknown or Not Reported | 1
Mean Young Mania Rating Scale (YMRS) Score [Mean (Standard Deviation); unit: score on a scale] — The Young Mania Rating Scale (YMRS) consists of 7 items rated on a scale from 0 (symptoms not present) to 4 (symptoms extremely severe) and 4 items rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe).The YMRS score ranges from 0-60. Questions are asked about the last week. A higher score signifies more severe manic symptoms.
  score on a scale | 23.8 (5.7)
Mean Children's Depression Rating Scale (CDRS) Score [Mean (Standard Deviation); unit: score on a scale] — The Children's Depression Rating Scale (CDRS) is a clinician-rated instrument with 17 items scored on a 1 to 5 or 1 to 7 scale. A rating of 1 indicates normal, thus the minimum score is 17. The maximum score is 113. Scores of 20-30 suggest borderline depression. Scores of 40-60 indicate moderate depression.
  score on a scale | 37.1 (11.7)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the Young Mania Rating Scale (YMRS) Score
Description: The Young Mania Rating Scale (YMRS) consists of 7 items rated on a scale from 0 (symptoms not present) to 4 (symptoms extremely severe) and 4 items rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe).The YMRS score ranges from 0-60. Questions are asked about the last week. A higher score signifies more severe manic symptoms.
Time Frame: Baseline and Endpoint (12 weeks or last observation carried forward if dropped prior to week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment With NAC
Number analyzed (Participants) | 26
score on a scale | -8.1 (8.5)

2. Secondary Outcome: Mean Change in the Children's Depression Rating Scale (CDRS) Score
Description: The Children's Depression Rating Scale (CDRS) is a clinician-rated instrument with 17 items scored on a 1 to 5 or 1 to 7 scale. A rating of 1 indicates normal, thus the minimum score is 17. The maximum score is 113. Scores of 20-30 suggest borderline depression. Scores of 40-60 indicate moderate depression.
Time Frame: Baseline and Endpoint (12 weeks or last observation carried forward if dropped prior to week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment With NAC
Number analyzed (Participants) | 26
score on a scale | -5.2 (10.7)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Consistent with good clinical practice, safety will be monitored by each subject's study clinician at each study visit. Subjects will be monitored by the study clinician for adverse events at each visit and adverse events will be recorded on an Adverse Events Form.
Arm/Group | Open-Label Treatment With NAC
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 2/29
Other Adverse Events (participants affected / at risk) | 17/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Treatment With NAC (N=29)
Hospitalization (Psychiatric disorders) | 1 (1)
Mania (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Treatment With NAC (N=29)
Nausea/Vomit/Diarrhea (Gastrointestinal disorders) | 7 (11)
Insomnia (Nervous system disorders) | 4 (4)
Cold/Infection/Allergy (Infections and infestations) | 4 (5)
Headache (General disorders) | 3 (3)
Anxious/Worried (Psychiatric disorders) | 2 (2)
Neurological (Nervous system disorders) | 2 (2)
Dizzy/Lightheaded (General disorders) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased Appetite (General disorders) | 1 (3)
Dermatological (Skin and subcutaneous tissue disorders) | 1 (2)
Thirsty (General disorders) | 1 (3)
Bike Injury (Stitches) (Injury, poisoning and procedural complications) | 1 (1)
Dissociation (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT02357290/Prot_SAP_000.pdf